CLINICAL TRIAL: NCT00053105
Title: A Phase I Trial of BBR 2778 in Combination With Cytarabine, Methylprednisolone and Cisplatin in the Treatment of Patients With Relapsed or Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy in Treating Patients With Relapsed or Refractory Aggressive Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000269140; THERADEX-AZA-I-05; NOVUSPHARMA-AZA-I-05; NOVUSPHARMA-AZA-1401; CWRU-050213J
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2003-03

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent grade 3 follicular lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, T-Cell, Cutaneous; Lymphoma, Large-Cell, Immunoblastic | interventions — Cisplatin; Cytarabine; Methylprednisolone

INTERVENTIONS:
Drug: cisplatin
Drug: cytarabine
Drug: methylprednisolone
Drug: pixantrone dimaleate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effect of combination chemotherapy on the body when treating patients who have relapsed or refractory aggressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended dose of pixantrone when administered with cytarabine, methylprednisolone, and cisplatin in patients with relapsed or refractory aggressive non-Hodgkin's lymphoma.
* Determine the dose-limiting toxic effects of this regimen in these patients.
* Determine the relationship between toxicity and systemic exposure to this regimen in these patients.
* Determine the safety of this regimen in these patients.
* Assess the pharmacokinetics of this regimen in these patients.
* Determine, preliminarily, the efficacy of this regimen in these patients.

OUTLINE: This is an open-label, non-randomized, multicenter, dose-escalation study of pixantrone.

Patients receive pixantrone IV over 1 hour on day 1, methylprednisolone IV over 15 minutes on days 1-5, cisplatin IV over 30 minutes on days 1-4, and cytarabine IV over 2 hours on day 5. Treatment repeats every 21 days for at least 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of pixantrone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 6 patients experience dose-limiting toxicity. Additional patients are treated at the recommended dose, which is defined as the dose preceding the MTD.

Patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 3-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed relapsed or refractory aggressive non-Hodgkin's lymphoma (NHL) including the following:

  * Diffuse large B-cell lymphoma
  * Transformed NHL
  * Follicular large cell lymphoma
  * Peripheral T-cell lymphoma
  * Unclassified aggressive histology (immunoblastic lymphoma)
* Must have received 1 to 3 prior chemotherapy treatment regimens (may include doxorubicin up to a cumulative dose of no greater than 450 mg/m^2)
* No Burkitt's lymphoma, lymphoblastic lymphoma, or mantle cell lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 to 64

Performance status

* WHO 0-1

Life expectancy

* At least 3 months

Hematopoietic

* Neutrophil count at least 1,500/mm^3*
* Platelet count at least 100,000/mm^3* NOTE: *Lower values may be accepted if evidence of bone marrow involvement

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)**
* Alkaline phosphatase no greater than 2 times ULN**
* AST or ALT no greater than 2 times ULN**
* No history or clinical symptoms of hepatitis B or C virus NOTE: **Higher values may be accepted if evidence of liver involvement

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* LVEF at least 50% by MUGA
* No clinically significant cardiovascular abnormalities
* No New York Heart Association class II-IV heart disease
* No myocardial infarction within the past 6 months
* No severe arrhythmia
* No uncontrolled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after study
* No history or clinical symptoms of HIV
* No clinically significant neurological abnormalities
* No serious uncontrolled infection (NCI CTC grade 3-4)
* No condition that would place the patient at undue risk or interfere with the study results

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior radioimmunotherapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* At least 1 year since prior platinum or cytarabine (unless complete response to treatment)
* At least 2 years since prior fludarabine or nitrosoureas
* No prior cumulative cisplatin greater than 600 mg/m^2

Endocrine therapy

* Not specified

Radiotherapy

* See Biologic therapy
* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to the whole pelvis

Surgery

* At least 1 week since prior minor surgery and recovered
* At least 4 weeks since prior major thoracic and/or abdominal surgery and recovered

Other

* At least 1 month since prior investigational drugs
* Recovered from prior therapy
* No other concurrent investigational drugs

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2002-02

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fayad, MD, Study Chair — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Ireland Cancer Center, Cleveland, Ohio
  - Boston Baskin Cancer Group, University Tennessee, Memphis, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas